CLINICAL TRIAL: NCT01003392
Title: Study of Coffee and Its Influence on the Heart in Normal People, Those With Coronary Artery Disease and Diabetics.
Brief Title: Influence of Coffee on the Health and on the Heart of Normal, Diabetics e Coronary Artery Disease Patients
Acronym: Coffee&Heart
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Feculdade de Medicina da Universidade de Sao Paulo - Brasil (Other)
Responsible Party: Principal Investigator, Luiz Antonio M. Cesar, Professor of Medicine, University of Sao Paulo
Other Study IDs: SDC2500/04/120; CAPPesq-879/04 (Other: CAPPesq)
Record Dates: First submitted 2009-10-26; First posted 2009-10-28 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Coffee; Heart system
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Normal: Normal volunteers, with no diagnosed chronic disease.
- Coronary artery disease: Group of patients with diagnosed coronary artery disease.
- Diabetes: Diabetic patients.

SUMMARY:
Coffee is a worldwide drink, been part of any culture. There are some concerns about effects of coffee on the health. Recently, epidemiological studies have shown benefits of coffee drinking to diabetics and also to prevent diabetes in populations. We aim to understand some effects of coffee and not only caffeine over vascular system, in special coronary artery disease patients, diabetics end normal people.

DETAILED DESCRIPTION:
Patients will have a wash-out period (21 days) with no coffee or other caffeine-drinks. Then they will be submitted to treadmill test, MAPA, Holter-ECG and vascular reactivity study, biochemical and inflammatory plasma dosages, as basal. Then they will start a period of coffee drinking over 4 weeks; and all exams will be repeated. We will study two types of coffee, arabica and robusta; with two types of toasted beans(regular and soft). Also regular and decaffeinated coffee. A total of 300 (100 normal people, 100 diabetics, 100 coronary disease) individuals will be tested.

ELIGIBILITY:
Inclusion Criteria:

Normal Volunteers:

1. Healthy volunteer.
2. Age between 20 and 80 years.
3. No addict to drugs.
4. Absence of chronicle diseases.
5. No alcohol abuse.
6. No smoker.

Coronary artery disease:

1. Presence of coronary artery disease, by coronary angiography
2. Stable angina, class 1-3 of CCS.
3. Age between 20 and 80 years.
4. Treadmill effort test with ischemia.
5. No alcohol abuse.
6. No smoker.

Diabetes:

1. Presence of type II Diabetes on oral treatment.
2. Age between 20 and 80 years.
3. Absence of chronicle diseases, except diabetes.
4. No alcohol abuse.
5. No smoker.

Exclusion Criteria:

Normal Volunteers:

1. Any blood test with twice or more the upper limit range.
2. Presence of enlarged QRS.

Coronary artery disease:

1. Any blood test with twice or more the upper limit range even with treatment.
2. Presence of enlarged QRS.
3. Ventricular dysfunction (EF < 45%).

Diabetes:

1. Blood glucose greater than 160 mg/dL.
2. Others blood tests with twice or more the upper limit range even with treatment.
3. Presence of enlarged QRS.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group of normal patients, group of patients with diagnosed coronary artery disease and group of diabetic patients.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2008-03; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Verify the relationship between coffee ingestion and cardiovascular morbidity and mortality | 10 years of follow-up

SECONDARY OUTCOMES:
Relationship between coffee ingestion and cardiovascular risk factors | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Luiz A Machado Cesar, PhD, MD., Study Chair — Heart Institute
Locations (1):
- Heart Institute (InCor), Univ. of Sao Paulo Medical School, São Paulo, São Paulo, Brazil